CLINICAL TRIAL: NCT03289520
Title: Effect of Clopidogrel on Early Failure of Arteriovenous Fistulas for Hemodialysis
Brief Title: Clopidogrel Prevention of Early Arteriovenous (AV) Fistula Thrombosis
Acronym: FISTULA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The Cleveland Clinic (Other); Boston University (Other); Duke University (Other); University of Iowa (Other); MaineHealth (Other); University of Texas Southwestern Medical Center (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other); Baystate Medical Center (Other); Vanderbilt University (Other); CAMC Health System (Other); Emory University (Other); St. Louis University (Other); Tyler Nephrology Associates (Unknown); Vascular Surgery Associates LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAC Fistula; U01DK058982 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Kidney Failure; Hemodialysis Fistula Thrombosis
Keywords: Access Blood Flow Monitoring; Clinical Trial Vascular Access; Fistula Failure; Hemodialysis; Vascular Access
MeSH Terms: conditions — Renal Insufficiency | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clopidogrel (Experimental)
  Interventions: Drug: Clopidogrel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clopidogrel
  Arms: Clopidogrel
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine whether clopidogrel reduces the early failure rate of native AV fistulae. This study was originally registered as NCT00067119 which included two protocols, this one and the GRAFT study)

ELIGIBILITY:
Fistula Study Protocol

Inclusion Criteria:

* Age 18-21 depending on state regulations
* Life expectancy of at least six months
* Chronic renal failure with anticipated start of hemodialysis within six months of enrollment, or current dialysis dependence
* Planned creation of native upper extremity AV fistula
* The patient is not on aspirin, or the patient is on aspirin but has not had a myocardial infarction or a cerebrovascular accident within the past 12 months.
* The patient is expected to stay at a participating dialysis facility for at least 6 months.
* The patient's physician(s) will allow the patient to participate.
* Ability to give informed consent.

Exclusion Criteria:

* Women must not be pregnant, breastfeeding, or plan to be pregnant during the course of the study.
* The presence of ongoing bleeding.
* The presence of a known bleeding disorder (e.g., hemophilia or von Willebrand's disease).
* Recent bleeding episode requiring transfusion within 12 weeks of entry.
* The presence of acute ulcer disease. Acute ulcer disease is defined as a new diagnosis of peptic disease including esophagitis, gastritis, or ulcer or the initiation of treatment with proton pump inhibitors, H2 blockers or therapy for Helicobacter pylori within three months prior to obtaining consent.
* A condition which prohibits discontinuation of anticoagulant drugs, aspirin, or nonsteroidal anti-inflammatory drugs during the six week study drug administration period. Use of heparin during dialysis is allowed.
* Required use of oral or intravenous glucocorticoids at a dose greater than the equivalent of prednisone 15 mg per day during the six week study drug administration period.
* Current unstable angina.
* Required use of clopidogrel.
* Known hypersensitivity to clopidogrel.
* Medical considerations making anti-platelet therapy dangerous.
* Current uncontrolled hypertension with systolic blood pressure in excess of 200 mm Hg or diastolic blood pressure in excess of 115 mm Hg at the time of enrollment.
* Baseline platelet count less than 75,000/mm3.
* Known advanced liver disease with decompensated cirrhosis, jaundice, ascites or bleeding varices.
* Current problem with substance abuse.
* Concurrent participation in another medical intervention trial.
* Anticipated non-compliance with medical care based on physician judgment.
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2003-01-07 (Actual); Primary Completion 2007-06-18 (Actual); Study Completion 2007-06-18 (Actual)

PRIMARY OUTCOMES:
Fistula thrombosis (patency failure) | 6 weeks
  The fistula was classified as patent if a bruit was audible with a stethoscope throughout systole and diastole at least 8 cm proximal to the arteriovenous anastomosis. Fistula patency was assessed by trained study personnel.

SECONDARY OUTCOMES:
Failure to attain suitability for dialysis (ability to use the fistula for dialysis with 2 needles and maintain a dialysis machine blood flow rate adequate for optimal dialysis (>=300 mL/min)) | 30 days
  Fistula suitability was defined as the ability to use the fistula for dialysis with 2 needles and maintain a dialysis machine blood flow rate adequate for optimal dialysis (>=300 mL/min) during 8 of 12 dialysis sessions occurring during a 30-day suitability ascertainment period. For participants receiving maintenance hemodialysis at the time of enrollment and for participants who started maintenance hemodialysis within 120 days after fistula creation, the suitability ascertainment period began between 120 and 150 days after fistula creation surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John W Kusek, Ph.D., Study Director — NIDDK - Telephone: 301-594-7717; Email: kusekj@ep.niddk.nih.gov; Catherine Meyers, M.D., Study Director — NIDDK - Telephone: 301-451-4901; Email: meyersc@extra.niddk.nih.gov
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Boston University Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository
Supporting Information: Study Protocol, SAP, CSR
URL: https://repository.niddk.nih.gov/study/84

REFERENCES:
- [Background] Dember LM, Kaufman JS, Beck GJ, Dixon BS, Gassman JJ, Greene T, Himmelfarb J, Hunsicker LG, Kusek JW, Lawson JH, Middleton JP, Radeva M, Schwab SJ, Whiting JF, Feldman HI; DAC Study Group. Design of the Dialysis Access Consortium (DAC) Clopidogrel Prevention of Early AV Fistula Thrombosis Trial. Clin Trials. 2005;2(5):413-22. doi: 10.1191/1740774505cn118oa. PMID 16317810
- [Result] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730